CLINICAL TRIAL: NCT05863195
Title: A Randomized Phase III Study of Systemic Therapy With or Without Hepatic Arterial Infusion for Unresectable Colorectal Liver Metastases: The PUMP Trial
Brief Title: Testing Pump Chemotherapy in Addition to Standard of Care Chemotherapy Versus Standard of Care Chemotherapy Alone for Patients With Unresectable Colorectal Liver Metastases: The PUMP Trial
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: ECOG-ACRIN Cancer Research Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Eastern Cooperative Oncology Group (Network)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EA2222; NCI-2023-02357 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EA2222 (Other: ECOG-ACRIN Cancer Research Group); EA2222 (Other: CTEP); U10CA180820 (NIH)
Record Dates: First submitted 2023-05-09; First posted 2023-05-17 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Colorectal Carcinoma; Metastatic Malignant Neoplasm in the Liver; Stage IV Colorectal Cancer AJCC v8; Unresectable Colorectal Carcinoma
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Bevacizumab; Immunoglobulin G; Disulfides; Cetuximab; Floxuridine; 5-fluoro-2'-deoxyuridine; Fluorouracil; dehydroftorafur; Drug Implants; Irinotecan; Leucovorin; Oxaliplatin; Panitumumab; X-Rays; Photons

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm A (HAI, floxuridine, standard chemotherapy) (Experimental): Patients undergo surgery to place the HAI pump, followed by SPECT/CT on study. Patients then receive floxuridine via the HAI pump on study. Patients also receive one of the following standard chemotherapy regimens per the treating physician: FOLFOX, FOLFIRI, or OX/IRI with or without cetuximab IV and/or panitumumab IV on study. Patients also undergo CT scans throughout the trial.
  Interventions: Biological: Cetuximab; Procedure: Computed Tomography; Drug: Floxuridine; Drug: Fluorouracil; Procedure: Implantation; Procedure: Intrahepatic Infusion Procedure; Drug: Irinotecan; Drug: Leucovorin; Drug: Oxaliplatin; Biological: Panitumumab; Procedure: Single Photon Emission Computed Tomography
- Arm B (standard chemotherapy) (Active Comparator): Patients receive one of the following standard chemotherapy regimens per the treating physician: FOLFOXIRI, FOLFOX, FOLFIRI, or OX/IRI with or without cetuximab IV, panitumumab IV, and/or bevacizumab IV on study. Patients also undergo CT scans throughout the trial.
  Interventions: Biological: Bevacizumab; Biological: Cetuximab; Procedure: Computed Tomography; Drug: Fluorouracil; Drug: Irinotecan; Drug: Leucovorin; Drug: Oxaliplatin; Biological: Panitumumab

INTERVENTIONS:
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Zirabev
  Arms: Arm B (standard chemotherapy)
Biological: Cetuximab — Given IV
  Other Names: Cetuximab Biosimilar CDP-1; Cetuximab Biosimilar CMAB009; Cetuximab Biosimilar KL 140; Chimeric Anti-EGFR Monoclonal Antibody; Chimeric MoAb C225; Chimeric Monoclonal Antibody C225; Erbitux; IMC-C225
Procedure: Computed Tomography — Undergo SPECT/CT and/or CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; CT; CT Scan; tomography
Drug: Floxuridine — Given via HAI pump
  Other Names: 2'-Deoxy-5-fluorouridine; 5-Fluoro-2'-deoxyuridine; 5-Fluorodeoxyuridine; 5-Fluorouracil deoxyriboside; 5-FUdR; FDUR; Floxuridin; Fluorodeoxyuridine; Fluorouridine Deoxyribose; Fluoruridine Deoxyribose; FUdR; WR-138720
  Arms: Arm A (HAI, floxuridine, standard chemotherapy)
Drug: Fluorouracil — Given IV
  Other Names: 5 Fluorouracil; 5 Fluorouracilum; 5 FU; 5-Fluoro-2,4(1H, 3H)-pyrimidinedione; 5-Fluorouracil; 5-Fluracil; 5-Fu; 5FU; AccuSite; Carac; Fluoro Uracil; Fluouracil; Flurablastin; Fluracedyl; Fluracil; Fluril; Fluroblastin; Ribofluor; Ro 2-9757; Ro-2-9757
Procedure: Implantation — Undergo surgery to place the HAI pump
  Arms: Arm A (HAI, floxuridine, standard chemotherapy)
Procedure: Intrahepatic Infusion Procedure — Undergo HAI
  Other Names: HAI; Hepatic Arterial Infusion; Hepatic Artery Infusion; IHI; Intrahepatic Infusion
  Arms: Arm A (HAI, floxuridine, standard chemotherapy)
Drug: Irinotecan — Given IV
Drug: Leucovorin — Given IV
  Other Names: Folinic acid
Drug: Oxaliplatin — Given IV
  Other Names: 1-OHP; Ai Heng; Aiheng; Dacotin; Dacplat; Diaminocyclohexane Oxalatoplatinum; Eloxatin; Eloxatine; JM-83; Oxalatoplatin; Oxalatoplatinum; RP 54780; RP-54780; SR-96669
Biological: Panitumumab — Given IV
  Other Names: ABX-EGF; ABX-EGF Monoclonal Antibody; ABX-EGF, Clone E7.6.3; E7.6.3; Human IgG2K Monoclonal Antibody; MoAb ABX-EGF; MoAb E7.6.3; Monoclonal Antibody ABX-EGF; Monoclonal Antibody E7.6.3; Vectibix
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
  Arms: Arm A (HAI, floxuridine, standard chemotherapy)

SUMMARY:
This phase III trial compares hepatic arterial infusion (HAI) (pump chemotherapy) in addition to standard of care chemotherapy versus standard of care chemotherapy alone in treating patients with colorectal cancer that has spread to the liver (liver metastases) and cannot be removed by surgery (unresectable). HAI uses a catheter to carry a tumor-killing chemotherapy drug called floxuridine directly into the liver. HAI is already approved by the Food and Drug Administration (FDA) for use in metastatic colorectal cancer to the liver, but it is only available at a small number of hospitals, and most of the time it is not used until standard chemotherapy stops working. Standard chemotherapy drugs work in different ways to stop the growth of tumor cells, either by killing the cells, by stopping them from dividing, or by stopping them from spreading. Adding HAI to standard chemotherapy may be effective in shrinking or stabilizing unresectable colorectal liver metastases.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To determine if patients with persistently unresectable colorectal liver metastases (CRLM) after treatment with first-line chemotherapy have improved overall survival (OS) with hepatic arterial infusion (HAI) and systemic chemotherapy versus systemic chemotherapy alone.

SECONDARY OBJECTIVES:

I. To determine whether there is a direct association between hepatic progression free survival (hPFS) and overall survival (OS) when patients are treated with HAI combined with systemic chemotherapy for unresectable CRLM.

II To determine the impact on progression free survival (overall, hepatic and extrahepatic) for patients with unresectable CRLM treated with HAI in combination with systemic chemotherapy.

III. To determine objective response rate (ORR) in the liver, defined as the proportion of patients achieving complete or partial response by Response Evaluation Criteria is Solid Tumors (RECIST) 1.1.

IV. To determine the rate of conversion to resectable disease, defined as the proportion of patients who successfully convert from unresectable to resectable status and undergo R0/R1 resection/ablation.

V. To determine the rate in which patients are intended to be treated with HAI but are deemed ineligible at the time of planned pump insertion due to detection of occult extrahepatic disease or unsuitable arterial anatomy (Intra-Operative Ineligibility, IOI).

VI. To determine the extent to which patient and disease-specific factors correlate with short- and long-term risk of HAI-specific complications.

OUTLINE: Patients are randomized to 1 of 2 arms.

ARM A: Patients undergo surgery to place the HAI pump, followed by single photon emission computed tomography/computed tomography (SPECT/CT) on study. Patients then receive floxuridine via the HAI pump on study. Patients also receive one of the following standard chemotherapy regimens per the treating physician: FOLFOX (fluorouracil intravenously [IV], oxaliplatin IV, and leucovorin IV), FOLFIRI (fluorouracil IV, irinotecan IV, and leucovorin IV), or OX/IRI (oxaliplatin IV and irinotecan IV) with or without cetuximab IV and/or panitumumab IV on study. Patients also undergo CT scans throughout the trial.

ARM B: Patients receive one of the following standard chemotherapy regimens per the treating physician: FOLFOXIRI (fluorouracil IV, oxaliplatin IV, irinotecan IV, and leucovorin IV), FOLFOX, FOLFIRI, or OX/IRI with or without cetuximab IV, panitumumab IV, and/or bevacizumab IV on study. Patients also undergo CT scans throughout the trial.

ELIGIBILITY:
Inclusion Criteria:

* Patient must be >= 18 years of age
* Patient must have confirmed unresectable liver confined metastatic colorectal cancer (CRC).

  * Patient must not have radiographically or clinically evident extrahepatic disease (including but not limited to radiographically positive periportal lymph nodes).

    * NOTE: Patients found to have positive periportal nodes at the time of HAI placement can remain on study.
  * Patient may have calcified pulmonary nodules, and/or =< 5 indeterminate and stable (for a minimum of 3 months on chemotherapy) pulmonary nodules each measuring =< 6 mm in maximal axial dimension.
  * Patient's primary tumor may be in place.
* Patient must have received 3-6 months of previous first-line chemotherapy that meet one of the following three criteria: a) have received at least 6 but no more than 12 cycles of first-line cytotoxic chemotherapy (where 1 cycle = 14 days) OR b) have received at least 4 but no more than 8 cycles of first-line cytotoxic chemotherapy (where 1 cycle = 21 days) OR c) have developed new colorectal liver metastases (CRLM) within 12 months of completing adjuvant systemic therapy for stage II-III colorectal cancer.

  * NOTE: First-line chemotherapy may have included any of the following regimens as listed in the National Comprehensive Cancer Network (NCCN) Guidelines: leucovorin calcium (folinic acid), fluorouracil, and oxaliplatin (FOLFOX) (or equivalent), leucovorin calcium (calcium folinate), 5-fluorouracil, and irinotecan (FOLFIRI) (or equivalent), leucovorin calcium (calcium folinate), 5-fluorouracil, oxaliplatin, and irinotecan (FOLFOXIRI), each with or without any of the following: bevacizumab, cetuximab, or panitumumab.
* Patient must have stable or responding disease on first-line chemotherapy by RECIST 1.1 criteria
* Patient must meet the following criteria for technical unresectability:

  * A margin-negative resection requires resection of three hepatic veins, both portal veins, or the retrohepatic vena cava OR a resection that leaves less than two adequately perfused and drained segments.
  * NOTE: Institutional multidisciplinary review is required to confirm unresectability and rule out radiographically positive extrahepatic disease.
* Patient must undergo CT angiography (chest/abdomen/pelvis) to confirm acceptable hepatic arterial anatomy for HAI and to rule out extrahepatic disease within 4 weeks prior to randomization.
* Patient must have an Eastern Cooperative Oncology Group (ECOG) Performance Status 0-1 and be clinically fit to undergo surgery as determined by the pre-operative evaluation.
* Leukocytes >= 3,000/mcL (obtained =< 14 days prior to protocol randomization)
* Absolute neutrophil count (ANC) >= 1,500/mcL (obtained =< 14 days prior to protocol randomization)
* Platelets >= 100,000/mcL (obtained =< 14 days prior to protocol randomization)
* Total Bilirubin =< 1.5 mg/dL (obtained =< 14 days prior to protocol randomization)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) =< 3.0 x institutional upper limit of normal (ULN) (obtained =< 14 days prior to protocol randomization)
* Creatinine =< 1.5 x institutional ULN OR creatinine clearance >= 50 mL/min calculated by the Cockcroft-Gault method (obtained =< 14 days prior to protocol randomization)
* Calcium >= institutional lower limit of normal (LLN)
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial.
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months of randomization are eligible for this trial. Testing for HIV is not required for entry onto the study

Exclusion Criteria:

* Patient must not have a liver tumor burden exceeding 70% of total liver volume.
* Patient must not have had prior radiation to the liver (prior radiation therapy to the pelvis is acceptable if completed at least 2 weeks prior to randomization).
* Patient must not have had prior trans-arterial bland embolization, chemoembolization (TACE) or radioembolization (TARE).
* Patient must not have had prior treatment with HAI/floxuridine (FUDR)
* Patient must not have microsatellite instability-high (MSI-H) colorectal cancer.
* Patient must not have CRLM that could be resected with 2-stage hepatectomy, including associating liver partition and portal vein ligation (ALPPS).
* Patient must not have an active infection, serious or non-healing active wound, ulcer, or bone fracture.
* Patient must not have any serious medical problems which would preclude receiving the protocol treatment or would interfere with the cooperation with the requirements of this trial.
* Patient must not have cirrhosis and/or clinical or radiographic evidence of portal hypertension
* Patient must not be pregnant or breast-feeding due to the potential harm to an unborn fetus and possible risk for adverse events in nursing infants with the treatment regimens being used.

  * All patients of childbearing potential must have a blood test or urine study within 14 days prior to randomization to rule out pregnancy.
  * A patient of childbearing potential is defined as anyone, regardless of sexual orientation or whether they have undergone tubal ligation, who meets the following criteria: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy; or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months).
* Patient must not expect to conceive or father children by using accepted and effective method(s) of contraception or by abstaining from sexual intercourse for the duration of their participation in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 408 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2034-06-30 (Estimated)

PRIMARY OUTCOMES:
Overall survival (OS) | From randomization to death from any cause, assessed up to 5 years
  Patients still living will be censored at the date last known alive. OS will be evaluated using the Kaplan-Meier method, and arms will be compared via a stratified log rank test.

SECONDARY OUTCOMES:
Progression free survival (PFS) | From randomization to first observed disease progression at any site, or death from any cause, assessed up to 5 years
  Patients still living without disease progression will be censored at the date of last disease assessment. Disease progression will be based on findings from surveillance cross-sectional imaging of the chest/abdomen/pelvis every 3 months after randomization, defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1. Will be analyzed similarly to OS, but with and without stratification for sensitivity.
Hepatic PFS | From randomization to first observed disease progression in the liver, or death from any cause, assessed up to 5 years
  Patients still living without hepatic disease progression will be censored at the date of last disease assessment. Hepatic disease progression will be based on findings from surveillance cross-sectional imaging of the chest/abdomen/pelvis every 3 months after randomization, defined by RECIST 1.1.
Extrahepatic-PFS | From randomization to first observed disease progression outside of the liver, or death from any cause, assessed up to 5 years
  Patients still living without extrahepatic disease progression will be censored at the date of last disease assessment. Extrahepatic disease progression will be based on findings from surveillance cross-sectional imaging of the chest/abdomen/pelvis every 3 months after randomization, defined by RECIST 1.1.
Objective response rate | Up to 5 years
  Will assess hepatic disease burden specifically. Defined as the proportion of patients achieving complete or partial response by RECIST 1.1. Response will be based on surveillance cross-sectional imaging of the chest/abdomen/pelvis every 3 months (+/- 2 weeks) after initiation of treatment (Arm A = surgery, Arm B = cycle 1, day 1 of chemotherapy). Arms will be compared via a Pearson chi-square test. All rates will be reported with exact binomial 95% confidence intervals.
Rate of conversion to resectable disease | Up to 5 years
  Defined as the proportion of patients who successfully convert from unresectable to resectable status and undergo R0/R1 resection/ablation. All rates will be reported with exact binomial 95% confidence intervals.
Intra-operative ineligibility rate | Up to 5 years
  Defined as the proportion of patients intended to receive hepatic arterial infusion that do not undergo pump implantation due to intraoperative detection of occult extrahepatic disease or unsuitable hepatic arterial anatomy. All rates will be reported with exact binomial 95% confidence intervals.
Incidence of adverse events | Up to 5 years
  Defined according to the Common Terminology Criteria for Adverse Events.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Lidsky, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (39):
- United States (39):
  - University of Alabama at Birmingham Cancer Center, Birmingham, Alabama
  - UCHealth University of Colorado Hospital, Aurora, Colorado
  - UM Sylvester Comprehensive Cancer Center at Aventura, Aventura, Florida
  - UM Sylvester Comprehensive Cancer Center at Coral Gables, Coral Gables, Florida
  - UM Sylvester Comprehensive Cancer Center at Deerfield Beach, Deerfield Beach, Florida
  - UM Sylvester Comprehensive Cancer Center at Hollywood, Hollywood, Florida
  - University of Miami Miller School of Medicine-Sylvester Cancer Center, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Kendall, Miami, Florida
  - UM Sylvester Comprehensive Cancer Center at Plantation, Plantation, Florida
  - Emory University Hospital/Winship Cancer Institute, Atlanta, Georgia
  - University of Chicago Comprehensive Cancer Center, Chicago, Illinois
  - Memorial Hospital East, Shiloh, Illinois
  - IU Health North Hospital, Carmel, Indiana
  - Indiana University/Melvin and Bren Simon Cancer Center, Indianapolis, Indiana
  - University of Kentucky/Markey Cancer Center, Lexington, Kentucky
  - University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan
  - Corewell Health Grand Rapids Hospitals - Butterworth Hospital, Grand Rapids, Michigan
  - Mayo Clinic in Rochester, Rochester, Minnesota
  - Siteman Cancer Center at Saint Peters Hospital, City of Saint Peters, Missouri
  - Siteman Cancer Center at West County Hospital, Creve Coeur, Missouri
  - Washington University School of Medicine, St Louis, Missouri
  - Siteman Cancer Center-South County, St Louis, Missouri
  - Siteman Cancer Center at Christian Hospital, St Louis, Missouri
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, East White Plains, New York
  - Mount Sinai Hospital, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York
  - Duke University Medical Center, Durham, North Carolina
  - Case Western Reserve University, Cleveland, Ohio
  - Fox Chase Cancer Center, Philadelphia, Pennsylvania
  - Allegheny General Hospital, Pittsburgh, Pennsylvania
  - West Penn Hospital, Pittsburgh, Pennsylvania
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Parkland Memorial Hospital, Dallas, Texas
  - UT Southwestern/Simmons Cancer Center-Dallas, Dallas, Texas